CLINICAL TRIAL: NCT01897948
Title: The Effects of Feeding Different Levels of Docosahexaenoic Acid to Pre-School Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non-compliance
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: University of Kansas (Other); John Colombo, PhD, The University of Kansas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 6022
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Measurement of Docosahexaenoic Acid Levels in Pre-school Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk-based beverage with DHA at mid-level (Experimental)
  Interventions: Other: Milk-based beverage with DHA at mid level
- Milk-based beverage with DHA at high level (Experimental)
  Interventions: Other: Milk-based beverage with DHA at high level
- Milk-based beverage without DHA (Active Comparator)
  Interventions: Other: Milk-based beverage without DHA

INTERVENTIONS:
Other: Milk-based beverage without DHA
  Arms: Milk-based beverage without DHA
Other: Milk-based beverage with DHA at mid level
  Arms: Milk-based beverage with DHA at mid-level
Other: Milk-based beverage with DHA at high level
  Arms: Milk-based beverage with DHA at high level

SUMMARY:
This clinical trial will measure Docosahexaenic Acid (DHA) levels in the blood and evaluate the relation to cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child is 3 years of age ± 90 days
* Weight for length is within 10th to 90th percentile as plotted on WHO growth charts
* Parent/caregiver reports that child consumes at least 6 oz of cow milk or cow milk-based beverages on a daily basis
* Parent is willing to exclude sources of DHA from child's diet during the study
* Parent agrees not to give vitamins to child during the study
* English is the primary language in the home
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* Gestational age at birth ≤ 36 weeks
* History of neuro/psychiatric conditions
* History of underlying metabolic or chronic disease
* Child is ill, has used antihistamines or diagnosed with an infection at time of cognitive testing
* History of suspected or known cow milk protein intolerance
* Child's diet contains sources of supplemental DHA more than one time per week
* Child is from a multiple birth and the sibling(s) are living in the same household
* Child is enrolled in another interventional clinical research study
* Use of antihistamines within 12 hours of cognitive testing

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell phospholipid weight percent of Docosahexaenoic Acid | 6 months
Cognitive Measures - Executive Function, Language Development, and Behavior Assessment | 6 months

SECONDARY OUTCOMES:
Fatty Acid Desaturase (FADS) genotypes | Once
Plasma Vitamin D levels | 6 months
Iron levels in the blood | 6 months
Blood Pressure | 6 months
Heart Rate | 6 months
Height and Weight | 6 months
Recall of dietary intake at each study visit | 6 months
Parental Product Assessment Questionnaire completed at Study Visit 2 | once
Medically-confirmed adverse events collected throughout the study period | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, M.D., Study Director — Mead Johnson Nutrition
Locations (1):
- Universty of Kansas Medical Center, Kansas City, Kansas, United States